CLINICAL TRIAL: NCT02373748
Title: A Prospective, Single Site, Single-arm Study Designed to Evaluate the Performance of the BioGaming Device (YuGo) in the Support of Physical Rehabilitation
Brief Title: Performance of the BioGaming Device (YuGo) in the Support of Physical Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaming Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111CLD
Record Dates: First submitted 2015-02-17; First posted 2015-02-27 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Physical Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioGaming YuGo System (Experimental)
  Interventions: Device: BioGaming YuGo System

INTERVENTIONS:
Device: BioGaming YuGo System — Subjects will perform a customized training program predefined in the BioGaming YuGo system.

SUMMARY:
The purpose of this study is to evaluate the movements performed according to the BioGaming YuGo software, and verify that they are rehabilitation movements.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing to comply with protocol-specified evaluations
* Subject signed informed consent

Exclusion Criteria:

* Pregnant or nursing female subjects
* Surgical procedures or injuries to the extremities that could potentially affect physical functions
* Neurological and/or vestibular disease
* Cognitive impairment
* Subjects taking any prescribed drugs that could potentially affect physical function and balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of BioGaming YuGo activity movements which are clinician recognized rehabilitation movements. | Baseline procedure
  Activity movements are assessed by independent clinicians.

SECONDARY OUTCOMES:
Safety - Record of any adverse event | Baseline procedure
  Any adverse event occurring during the baseline procedure will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel